CLINICAL TRIAL: NCT03306160
Title: Prognostic Value of Central and BracHial Ambulatory Blood Pressure Monitoring in ERSD Patients Treated With HeMOdialysis: the C-HEMO Study
Brief Title: Prognostic Value of Central and BracHial Ambulatory Blood Pressure Monitoring in ERSD Patients Treated With HeMOdialysis
Acronym: C-HEMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, The chief director of department of cardiology, Shanghai 10th People's Hospital
Other Study IDs: C-HEMO001
Record Dates: First submitted 2017-09-28; First posted 2017-10-10 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: End Stage Renal Disease
Keywords: central blood pressure; ambulatory blood pressure monitoring; blood pressure variability
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: 48-hour blood pressure ambulatory monitoring — at first-time dialysis after enrollment, each patient will receive brachial and central blood pressure monitoring for 48 hours using a validate and commercially available device Mobil-O-Graph (IEM, Germany).

SUMMARY:
This is a prospective cohort study which aims to explore the significance of brachial and central ambulatory blood pressure monitoring in predicting cardiovascular risk in patients with end stage renal disease who are treated with hemodialysis. Enrolled patients will receive a 48-hour central and brachial ambulatory blood pressure monitoring at its first-time dialysis after enrollment. And their cardiovascular events and deaths at first and third year will be followed-up.

DETAILED DESCRIPTION:
The protocol of this study was approved by the local ethical review board. The including criteria: 1) ESRD treated with hemodialysis for more than 3 months prior to study enrollment; 2) agree to participate the study and sign informed written consent; 3) available for long-term follow-up. The excluding criteria: 1)chronic atrial fibrillation or other cardiac arrhythmia; 2) nonfunctional arteriovenous fistula in the contralateral brachial area of the one used for dialysis; 3) myocardial infarction, angina pectoris and ischemic stroke during the previous month; 4) congestive heart failure class IV based on the New York Heart Association classification; 5) malignancy or any other condition with poor prognosis; 6) antihypertensive treatment during one month prior to enrollment. After enrollment, every patient will receive a question-based interview to obtain medical history and the following examinations and tests: anthropometric parameters measurement including body height, weight; biochemical tests including vein blood and urine. At the first-time dialysis after enrollment, patients will receive 48-hour central and brachial ambulatory blood pressure monitoring using a well validated and commercial device Mobil-O-Graph (IEM, Germany). Brachial blood pressure are measured for each patient before every dialysis for at three month. Then one-year and three-year cardiovascular events and deaths will be followed-up. The primary outcome measures are as follows: deaths and cardiovascular events including nonfatal myocardial infarction, unstable angina, stroke, hospitalization for heart failure, or resuscitated cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage renal disease treated with hemodialysis for more than 3 months prior to study enrollment;
* agree to participate the study and sign informed written consent;
* available for long-term follow-up.

Exclusion Criteria:

* chronic atrial fibrillation or other cardiac arrhythmia;
* nonfunctional arteriovenous fistula in the contralateral brachial area of the one used for dialysis;
* myocardial infarction, angina pectoris and ischemic stroke during the previous month;
* congestive heart failure class IV based on the New York Heart Association classification;
* malignancy or any other condition with poor prognosis;
* antihypertensive treatment during 1 month prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with end-stage renal disease treated with hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-10-09 (Estimated); Study Completion 2020-10-09 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 3 year
  nonfatal myocardial infarction, unstable angina, stroke, hospitalization for heart failure, or resuscitated cardiac arrest
cardiovascular deaths | 3 year
  cardiovascular deaths
all-cause deaths | 3 year
  all-cause deaths

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, MD, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sumida K, Molnar MZ, Potukuchi PK, Thomas F, Lu JL, Yamagata K, Kalantar-Zadeh K, Kovesdy CP. Pre-end-stage renal disease visit-to-visit systolic blood pressure variability and post-end-stage renal disease mortality in incident dialysis patients. J Hypertens. 2017 Sep;35(9):1816-1824. doi: 10.1097/HJH.0000000000001376. PMID 28399042
- [Background] Karpetas A, Sarafidis PA, Georgianos PI, Protogerou A, Vakianis P, Koutroumpas G, Raptis V, Stamatiadis DN, Syrganis C, Liakopoulos V, Efstratiadis G, Lasaridis AN. Ambulatory recording of wave reflections and arterial stiffness during intra- and interdialytic periods in patients treated with dialysis. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):630-8. doi: 10.2215/CJN.08180814. Epub 2015 Jan 29. PMID 25635033
- [Background] Covic A, Goldsmith DJ, Panaghiu L, Covic M, Sedor J. Analysis of the effect of hemodialysis on peripheral and central arterial pressure waveforms. Kidney Int. 2000 Jun;57(6):2634-43. doi: 10.1046/j.1523-1755.2000.00124.x. PMID 10844634
- [Background] Ohno Y, Kanno Y, Takenaka T. Central blood pressure and chronic kidney disease. World J Nephrol. 2016 Jan 6;5(1):90-100. doi: 10.5527/wjn.v5.i1.90. PMID 26788468